CLINICAL TRIAL: NCT01102530
Title: Diabetes Prevention in Women With a Recent History of Gestational Diabetes
Brief Title: Diabetes Prevention in Women With a Recent History of Gestational Diabetes (Focus Groups)
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Sue E. Levkoff, ScD, Brigham and Women's Hospital
Other Study IDs: 2009p000042; MM-1094-09/09 (Other Grant/Funding Number: Center for Disease Control (CDC))
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this research is to conduct focus groups in order to adapt the Diabetes Prevention Program (DPP) so that it may successfully target women diagnosed with gestational diabetes (GDM) who are at high risk for developing Type 2 diabetes in the post-partum period. As this research seeks to gather formative data for a future intervention, the focus groups will: 1) provide information to maximize participation in the future intervention and 2) inform the location, content and format of the intervention.

We will be conducting focus groups and informant interviews to determine the DPP modifications necessary for adapting to the post-partum lifestyles of women with a recent history of GDM. Subjects will attend a 1 hour focus group or phone interview where they will be encouraged to respond to the facilitators' questions and to each other's comments on topics such as: gestational diabetes, healthy eating, exercise, and other type 2 diabetes prevention related activities. Working with a variety of health care providers, including endocrinologists, obstetricians and nurse-practitioners, we will identify and enroll up to 60 women total who are either current GDM patients at BWH or have a recent history of GDM who have delivered at Brigham and Women's Hospital in the last 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women ages 18-45
* Diagnosis of gestational diabetes within the past 5 years (Carpenter-Coustan criteria)
* English-speaking
* Currently not diagnosed with type 2 diabetes

Exclusion Criteria:

* Diagnosis of type 2 diabetes
* Non-English-speaking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy women with a diagnosis of gestational diabetes during a pregnancy within the past 5 years
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue E Levkoff, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Nicklas JM, Zera CA, Seely EW, Abdul-Rahim ZS, Rudloff ND, Levkoff SE. Identifying postpartum intervention approaches to prevent type 2 diabetes in women with a history of gestational diabetes. BMC Pregnancy Childbirth. 2011 Mar 24;11:23. doi: 10.1186/1471-2393-11-23. PMID 21435246